CLINICAL TRIAL: NCT06725316
Title: The Effect Of 4-7-8 Breathıng Exercıses on Paın, Vıtal Sıgns and Development ff Complıcatıons After Laparoscopıc Gynaecologıcal Surgery
Brief Title: The Effect Of 4-7-8 Breathıng Exercıs After Laparoscopıc Surgery
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Gazi University (Other)
Responsible Party: Principal Investigator, Canan Uçakçı Asalıoğlu, Principal Investigator, Gazi University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: CUA
Record Dates: First submitted 2024-10-10; First posted 2024-12-10 (Actual); Last update posted 2024-12-10 (Actual); Status verified 2024-12

CONDITIONS: Pain
Keywords: 4-7-8 breathing exercises; gynaecological surgery; pain; complication; vital signs
MeSH Terms: conditions — Pain

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- control group (No Intervention): Women in the control group will receive routine care in the hospital. Vital signs assessment form will be used to evaluate vital signs and development of complications in the first 8 hours of the postoperative period. The 'Mcgill Pain Scale Short Form' form will be used to evaluate the pain of the patients and the pain of the patient will be evaluated 4 times in total, at two, four, six and eight hours post-op.
- Experimental Group (Experimental): The women in the experimental group will be taught 4-7-8 breathing exercises before the operation. After making sure that they perform these exercises correctly, the training will be terminated. In order to perform the 4-7-8 exercise correctly and easily, an audible second counting application will be installed on the participants' phones and an hourly reminder alarm will be set. Participants will perform the first exercise with the postoperative nurse and the following exercises by themselves. Participants will be asked to do the exercise four times every hour for the first 8 hours postoperatively.
  Vital signs assessment form will be used to evaluate vital signs and development of complications in the first 8 hours postoperatively. The 'Mcgill Pain Scale Short Form' form will be used to evaluate the pain of the patients and the patient's pain will be evaluated 4 times in total, at two, four, six and eight hours post-op.
  Interventions: Behavioral: 4-7-8 breathing exercises

INTERVENTIONS:
Behavioral: 4-7-8 breathing exercises — Steps of doing 4-7-8 breathing exercise; firstly, the breath taken is exhaled completely through the mouth as if whistling. Then the lips are closed and inhaled quietly through the nose (4 seconds). The breath is held for seven seconds. At the last stage, the lips are tightened and exhaled through the mouth for 8 seconds. Then normal breathing is done for one minute. Breathing is repeated four times every hour.
  Arms: Experimental Group

SUMMARY:
The study was a single-centre, parallel randomised controlled experimental study conducted with block randomisation method.

DETAILED DESCRIPTION:
In determining the sample of the research, power analysis was performed and it was planned to have a total of 62 participants, with 31 participants in each group.Women undergoing gynaecological operations will be recruited in the order of hospitalisation according to the block randomisation method. The letters A and B in the blocks will be determined as experimental or control according to the coin flip method. One of the researchers will evaluate the participants according to the inclusion criteria and randomly assign them according to the block order after obtaining their informed consent. One of the researchers in this study will carry out the application. The other researchers will be blinded. The data obtained will be analysed by an independent statistician. Participant blinding will not be performed since the participants were informed about the study in informed consent. Descriptive Information Form, Mcgill Pain Scale Short Form (Biçici, 2010) and Vital Signs Assessment Form to evaluate vital signs and mobilisation will be used for data collection.Women who applied to the hospital due to benign gynaecological disorders and underwent laparoscopic surgery will first be evaluated whether they are eligible for the study according to the inclusion criteria evaluation form. Afterwards, women who are eligible to participate in the study will be randomly assigned by an independent researcher to determine whether they are in the experimental or control group.

ELIGIBILITY:
Inclusion Criteria:

Being literate, Having benign gynaecological disease, Not having any other disease affecting pain/living findings (neuropathy, migraine, Cardiovascular diseases, oncological disease, ...), Not using painkillers regularly, Not having substance addiction, Not having communication barrier.

Exclusion Criteria:

It was determined that women did not perform 4-7-8 breathing exercises regularly, Women wanted to leave the study, Complications related to surgery occurred at any stage of the study, Women did not complete the data collection tools.

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 62 (Estimated)
Dates: Start 2024-11-30 (Estimated); Primary Completion 2025-03-30 (Estimated); Study Completion 2025-03-30 (Estimated)

PRIMARY OUTCOMES:
vital signs assessment form | post-op will be evaluated 4 times in total, at two, four, six, eight hours.
  It was created by the researchers and will be used to determine blood pressure, pulse rate, painkiller use and complication development status.
Mcgill Pain Scale Short Form | post-op will be evaluated 4 times in total, at two, four, six, eight hours.
  The Short Form of the McGill Pain Scale consists of three parts.As the scores increase in this scale, it is seen that the pain level increases.